CLINICAL TRIAL: NCT06078033
Title: Efficacy of Mobilization With Movement on Conditioned Pain Modulation in Chronic Low Back Pain Patients: A Randomized Controlled Trial
Brief Title: Efficacy of Mobilization With Movement on Conditioned Pain Modulation in Chronic Low Back Pain Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Eleuterio Atanasio Sánchez Romero (Other)
Responsible Party: Sponsor-Investigator, Eleuterio Atanasio Sánchez Romero, PhD, Clinical Professor, Universidad Europea de Madrid
Organization: Universidad Europea de Madrid (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 1811202225222
Record Dates: First submitted 2023-09-29; First posted 2023-10-11 (Actual); Last update posted 2024-05-21 (Actual); Status verified 2024-05

CONDITIONS: Chronic Low-back Pain
Keywords: Chronic low back pain; Manual therapy; Conditioned Pain Modulation
MeSH Terms: interventions — Movement

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Masking Description: Randomization was conducted by single randomization. Allocation of the selected patients to different groups (A, intervention; B, placebo) was implemented by opaque envelopes. The randomization was performed by personnel not involved in the trial, such as clinics receptionist. The personnel placed the random characters into sealed opaque envelopes and provided the group allocation to patients. The envelopes were opened only by the manual therapist, without letting the patient know to which group they were assigned to. Additionally, outcomes assessor was blinded to which group patients were assigned to.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention: Mobilization with movement (MWM) (Experimental): The MWM technique was performed by asking patients to perform their painful movement (flexion, extension…). If pain was not reproduced, a combination of movements (flexion + rotation…) was performed. The most painful vertebral level was also evaluated with passive accessory vertebral movements. Then, with the patient in a seated position on a stretcher with the feet supported and a belt around the waist, the therapist performed a sustained glide over the targeted vertebra (spinous process) with the force and direction that relieved pain to the lowest level and asked the patient to perform his previous painful movement, as described by Mulligan. Three sets of 10 repetitions were performed, with 1-2 minutes rest between sets.
  Interventions: Biological: Mobilization with movement
- Control: Sham mobilization with movement (Sham Comparator): Patients allocated to sham group received same evaluation and treatment process. However, only manual contact was performed over the spinous process of the targeted vertebra, without the sustained glide and without applying any force. Three sets of 10 repetitions were performed, with 1-2 minutes rest between sets.
  Interventions: Biological: Sham mobilization with movement

INTERVENTIONS:
Biological: Mobilization with movement — Sustained neutral apophyseal glide (SNAG) mobilization with movement applied to targeted vertebra while patients performed their painful movement.
  Arms: Intervention: Mobilization with movement (MWM)
Biological: Sham mobilization with movement — Manual contact (without any pressure) applied to targeted vertebra while patients performed their painful movement.
  Arms: Control: Sham mobilization with movement

SUMMARY:
Patients with chronic low back pain may have altered endogenous mechanisms, which can be evaluated with conditioned modulation paradigms. Mobilization with movement has demonstrated improvements in endogenous analgesic mechanisms in conditions such as knee osteoarthritis or lateral epicondylalgia. However, its effects have not yet been studied in patients with chronic low back pain. The objective of this randomized clinical trial is to evaluate the efficacy of mobilization with movement compared to placebo on endogenous mechanisms in patients with chronic low back pain.

DETAILED DESCRIPTION:
Low back pain is the leading cause of disability worldwide, and chronic low back pain (CLBP) has a prevalence of 2-25%, 80% of which are classified as non-specific low back pain because the causal factors have not yet been determined. Although different mechanisms can be attributed to the chronification of pain, a frequent denominator is the amplification of nociceptive transmission or decreased inhibition of nociceptive stimuli in the peripheral and/or central nervous system.

To assess inhibitory pathways, conditioned pain modulation (CPM) paradigms are commonly used in humans. They are based on the idea that a noxious stimulus applied to one part of the body can inhibit pain elsewhere by activating the descending inhibitory system.

When CPM is evaluated in patients with chronic low back pain, contradictory results are found, with studies reporting an alteration of pain modulation mechanisms and others not.

Different studies found that manual therapy can improve CPM compared to sham in patients with chronic musculoskeletal pain, such as lateral epicondylalgia or knee osteoarthritis. However, its effects in patients with chronic low back pain have not yet been studied.

Therefore, the aim of this study was to investigate the effect of mobilization with motion on CPM in patients with chronic musculoskeletal pain.

ELIGIBILITY:
Inclusion Criteria:

* Adults with chronic low back pain (>3 months of pain duration)
* 2 or more on a scale of 0 to 10.

Exclusion Criteria:

* Radiculopathy
* Neurological signs, symptoms, or deficit
* Rheumatic or autoimmune disease
* Cutaneous disease
* History of fracture or spinal surgery
* Pregnancy
* Neuropathic pain
* Active cancer
* Spondylolysis/Spondylolisthesis
* Mild/Severe cognitive impairment which interferes with outcomes measurement

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 58 (Actual)
Dates: Start 2023-12-02 (Actual); Primary Completion 2024-05-20 (Actual); Study Completion 2024-05-20 (Actual)

PRIMARY OUTCOMES:
Conditioned pain modulation | 30 minutes
  Conditioned pain modulation of low back, measured on interspace between L5 and S1. Pressure pain threshold (PPT) was used as test stimulus while ischemic pain (using cuff) was used as conditioning stimulus. CPM effect were calculated as the differences between the PPT values with and without the conditioning stimulus.

SECONDARY OUTCOMES:
Pressure pain threshold | 30 minutes
  Pressure pain thresholds (PPT), measured on interspace between L5 and S1. PPT were measured with an algometer placed and applied perpendicular to the skin. Pressure was gradually increased at a rate of 1kg/sec over the targeted location until patient indicated verbally that the sensation became painful. Measurements were taken two times at the location with 30 seconds rest interval between each measurement. The mean of the two measurements for targeted location was calculated for statistical analysis.
Body Chart | Baseline
  Widespread pain was measured with body chart
Kinesiophobia | Baseline
  Kinesiophobia was measured with Spanish version of Tampa Scale of Kinesiophobia. Higher scores denotes greater fear of experiencing pain while moving.
Depression | Baseline
  Depressive symptoms were measured with Spanish version of Beck Inventory II. 0-13 normal scores; 14-19 mild; 20-28 moderate; 29-63 severe depression.
Anxiety | Baseline
  Anxiety was measured with Spanish version of State-trait Anxiety Inventory (STAI). Scores of 20-37 indicate no or low anxiety; 38-44 moderate anxiety; 45-80 high anxiety.
Disability | Baseline
  Low back pain associated disability was measured with Spanish version of Roland-Morris Disability Questionnaire. Higher scores denotes greater pain-associated disability.
Quality of life (QoL) | Baseline
  QoL was measured with Spanish version of EuroQol 5-Dimensions. Quality of life visual analogue scale consist of a scale from 0 (worse quality of life) to 100 (best quality of life). Additionally, quality of life index may be summarised by a series of five sentences, one for each dimension and stating the level within that dimension; or a label consisting of five ordinal numbers, one for each dimension (by convention, in the order these appear in the questionnaire), defining the severity level, where 1 means no problems.

CONTACTS AND LOCATIONS:
Overall Officials: Oliver Martínez, PhDc, Principal Investigator — Universidad Europea de Madrid
Locations (1):
- Universidad Europea de Madrid, Villaviciosa de Odón, Madrid, Spain

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Martinez-Pozas O, Sanchez-Romero EA, Beltran-Alacreu H, Arribas-Romano A, Cuenca-Martinez F, Villafane JH, Fernandez-Carnero J. Effects of Orthopedic Manual Therapy on Pain Sensitization in Patients With Chronic Musculoskeletal Pain: An Umbrella Review With Meta-Meta-analysis. Am J Phys Med Rehabil. 2023 Oct 1;102(10):879-885. doi: 10.1097/PHM.0000000000002239. Epub 2023 Mar 14. PMID 36917046
- [Result] Aoyagi K, He J, Nicol AL, Clauw DJ, Kluding PM, Jernigan S, Sharma NK. A Subgroup of Chronic Low Back Pain Patients With Central Sensitization. Clin J Pain. 2019 Nov;35(11):869-879. doi: 10.1097/AJP.0000000000000755. PMID 31408011
- [Result] Sánchez-Romero EA, González-Zamorano Y, Arribas-Romano A, Martínez-Pozas O, Fernández Espinar E, Pedersini P, Villafañe JH, Alonso Pérez JL, Fernández-Carnero J. Efficacy of Manual Therapy on Facilitatory Nociception and Endogenous Pain Modulation in Older Adults with Knee Osteoarthritis: A Case Series. Applied Sciences. 2021; 11(4):1895. https://doi.org/10.3390/app11041895
- [Result] McPhee ME, Vaegter HB, Graven-Nielsen T. Alterations in pronociceptive and antinociceptive mechanisms in patients with low back pain: a systematic review with meta-analysis. Pain. 2020 Mar;161(3):464-475. doi: 10.1097/j.pain.0000000000001737. PMID 32049888
- [Result] Neelapala YVR, Bhagat M, Frey-Law L. Conditioned Pain Modulation in Chronic Low Back Pain: A Systematic Review of Literature. Clin J Pain. 2020 Feb;36(2):135-141. doi: 10.1097/AJP.0000000000000778. PMID 31764164
- [Result] den Bandt HL, Paulis WD, Beckwee D, Ickmans K, Nijs J, Voogt L. Pain Mechanisms in Low Back Pain: A Systematic Review With Meta-analysis of Mechanical Quantitative Sensory Testing Outcomes in People With Nonspecific Low Back Pain. J Orthop Sports Phys Ther. 2019 Oct;49(10):698-715. doi: 10.2519/jospt.2019.8876. Epub 2019 Aug 23. PMID 31443625
- [Result] Bisset L, Paungmali A, Vicenzino B, Beller E. A systematic review and meta-analysis of clinical trials on physical interventions for lateral epicondylalgia. Br J Sports Med. 2005 Jul;39(7):411-22; discussion 411-22. doi: 10.1136/bjsm.2004.016170. PMID 15976161